CLINICAL TRIAL: NCT02605642
Title: PERSIST: PROSPECTIVE OBSERVATIONAL COHORT STUDY TO ASSESS PERSISTENCE OF CT-P13 (INFLIXIMAB) IN PATIENTS WITH RHEUMATOID DISEASES WHO ARE EITHER NAIVE TO BIOLOGICS OR SWITCHED FROM STABLE REMICADE(R) (INFLIXIMAB)
Brief Title: Post-Marketing Use Of CT-P13 (Infliximab) For Standard Of Care Treatment Of Rheumatoid Diseases Who Are Naïve To Biologics Or Switched From Remicade
Acronym: PERSIST
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: ZOBINF1505; C1231002 (Other: Alias Study Number)
Record Dates: First submitted 2015-09-02; First posted 2015-11-16 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Rheumatoid Diseases; Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis
Keywords: CT-P13; Inflectra; Remsima; Remicade; Infliximab; Observational; Follow-up; Safety
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic | interventions — CT-P13; Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CT-P13: biosimilar infliximab
  Interventions: Drug: CT-P13

INTERVENTIONS:
Drug: CT-P13 — biosimilar infliximab
  Other Names: Inflectra; Remsima

SUMMARY:
To assess persistence of CT-P13 in patients with Rheumatoid Diseases (Rheumatoid arthritis [RA], ankylosing spondylitis [AS], and psoriatic arthritis [PsA]) who are naïve to biologics or are switching from stable Remicade to CT-P13. The main objectives of the study are:

* To evaluate real-life drug persistence in RA, AS, and PsA patients who are either initiated with CT-P13 as their first biologic, or who are switched from stable Remicade
* To characterise the patient populations and drug usage patterns of RA, AS, and PsA patients who are either initiated with CT-P13 as their first biologic, or who are switched from stable Remicade
* To assess the safety of CT-P13 in RA, AS, and PsA patients who are either initiated with CT-P13 as their first biologic, or who are switched from stable Remicade for up to 2 years

DETAILED DESCRIPTION:
The study will be conducted in accordance with legal and regulatory requirements with scientific purpose, value and rigor following generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP), Good Epidemiological Practice (GEP), Good Practices for Outcomes Research, International Ethical Guidelines for Epidemiological Research, European Medicines Agency (EMA) European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) Guide on Methodological Standards in Pharmacoepidemiology, and FDA Guidance for Industry. Data sources will be validated and will consist of the hospital medical records and monitoring will be organized on a regular basis. Data sources will be validated. The source data will consist of medical records, physician questionnaires, and patient questionnaires. Data for the study will be entered into an electronic data capture system. Questionnaires will be completed on electronic tablets. The study is a one year enrollment period with a two year follow-up period. The study plans to enroll patients throughout Canada and Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years old at the time of enrollment
2. Patients who are prescribed CT-P13 or Remicade for the treatment of rheumatoid arthritis, ankylosing spondylitis, and psoriatic arthritis prescribed according to the corresponding summary of product characteristics (SmPC and Product Monograph) as determined by the investigator

Exclusion Criteria:

1. Any reported contraindications for Inflectra according to the SmPC or Product Monograph
2. Known hypersensitivity (including severe, acute infusion reactions) to infliximab, its excipients or other murine proteins, at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will include biologic naïve rheumatoid arthritis, ankylosing spondylitis, and psoriatic arthritis patients starting biologic treatment with CT-P13 or those switched to CT-P13 from stable Remicade treatment
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- Bulgaria (3):
  - MHAT Trimontium OOD, Plovdiv
  - MHAT Kaspela EOOD, Plovdiv
  - Diagnostic Consultative Center 17 Sofia EOOD, Sofia
- Canada (17):
  - Lucere Skin Dermatology & Laser Clinic, Edmonton, Alberta
  - Nexus Clinical Research, St. John's, Newfoundland and Labrador
  - Dr. Juris Lazovskis Inc., Sydney, Nova Scotia
  - The Waterside Clinic, Barrie, Ontario
  - William Osler Health System, Brampton, Ontario
  - Adachi Medicine Professional Corporation, Hamilton, Ontario
  - K-W Musculoskeletal Research Inc, Kitchener, Ontario
  - Y. Liu Medicine Professional, Milton, Ontario
  - Credit Valley Imaging Associates, Mississauga, Ontario
  - Oakville Rheumatology & Osteoporosis, Oakville, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Arthur Karasik Medicine Professional Corporation, Toronto, Ontario
  - Dr. Sabeen Anwar Medicine Professional Corporation, Windsor, Ontario
  - Centre Hospitalier de l'Universite de Montreal - Notre-Dame Hospital, Montreal, Quebec
  - Groupe de Recherche en Rhumatologie et Maladies Osseuses (GRMO), Québec, Quebec
  - Centre Rhumatologie de l'Est, Rimouski, Quebec
  - Centre de Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Czechia (2):
  - Revmatolog Mudr. Sirova Klara s.r.o., Ostrava
  - Revmatologický Ústav (RÚ), Prague
- Germany (10):
  - Rheumapraxis Steglitz, Berlin
  - Immanuel Diakonie GmbH, Bernau
  - Rheumatologisches MVZ Dresden GmbH, Dresden
  - Asklepios Gesundheitszentrum Elmshorn, Elmshorn
  - Rheumatologische Praxis Dr. med. Kühne, Haldensleben I
  - Dr. med. Jörg Kaufmann, Ludwigsfelde
  - Praxis Dr. Herbert Kellner, München
  - MVZ für Rheumatologie Dr. Martin Welcker GmbH, Planegg
  - Berufsausübungsgemeinschaft Martin Bohl-Bühler & Dr. med. Sabine Reckert, Potsdam
  - Dr. med. Jochen Walter - FA für Innere Medizin Rheumatologe, Rendsburg
- University General Hospital of Heraklion, Heraklion, Crete, Greece
- Spain (3):
  - Complexo Hospitalario Universitario A Coruña, A Coruña A Coruña
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
- United Kingdom (2):
  - Portsmouth Hospitals NHS Trust - Queen Alexandra Hospital, Portsmouth
  - Salisbury NHS Foundation Trust - Salisbury District Hospital, Sailsbury

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Taylor PC, Christensen R, Moosavi S, Selema P, Guilatco R, Fowler H, Mueller M, Liau KF, Haraoui B. Real-life drug persistence in patients with rheumatic diseases treated with CT-P13: a prospective observational cohort study (PERSIST). Rheumatol Adv Pract. 2021 Apr 23;5(2):rkab026. doi: 10.1093/rap/rkab026. eCollection 2021. PMID 34377890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 351 participants were included in this study, however, 17 participants were excluded from all analysis (they were neither BDMARD naive nor switched from Remicade). They switched to CT-P13 from a BDMARD other than Remicade, therefore not considered for any analysis.
Groups:
- Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive: BDMARD naive participants who were receiving CT-P13 according to the summary of product characteristics (SmPC and Product Monograph) as determined by the investigator, were included in this group and observed in this study for a duration of up to 2 years.
- Participants Who Switched From Remicade to CT-P13: Participants who were previously treated with Remicade, switched to CT-P13 and started receiving CT-P13 (according to the SmPC and Product Monograph; as determined by the investigator) from stable treatment with Remicade, were included in this group and observed for a duration of up to 2 years.
Period: Overall Study
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Started | 227 | 107
Safety Set (Included all participants who received at least 1 dose of CT- P13 during study observation period) | 221 | 107
Completed | 131 | 86
Not Completed | 96 | 21
Not completed — Other | 11 | 1
Not completed — Participant non-compliance | 2 | 4
Not completed — Physician Decision | 10 | 0
Not completed — Lost to Follow-up | 12 | 1
Not completed — Adverse Event | 14 | 2
Not completed — Withdrawal by Subject | 23 | 2
Not completed — Lack of response | 24 | 11

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of CT-P13 during the study observation period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13 | Total
Number analyzed (Participants) | 221 | 107 | 328
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (13.54) | 52.5 (12.61) | 53.1 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 48 | 166
  Male | 103 | 59 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 212 | 106 | 318
  Black or African American | 2 | 0 | 2
  Asian | 6 | 0 | 6
  Other | 1 | 1 | 2
Height [Mean (Standard Deviation); unit: centimeter] — Population: Number analyzed signifies participants evaluable for this baseline measure.
  centimeter
    number analyzed (Participants) | 220 | 106 | 326
    (all) | 168.44 (9.467) | 173.19 (10.592) | 169.98 (10.080)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 80.80 (16.613) | 83.21 (19.442) | 81.59 (17.592)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per meter square] — Population: Number analyzed signifies participants evaluable for this baseline measure.
  kilogram per meter square
    number analyzed (Participants) | 220 | 106 | 326
    (all) | 28.51 (5.521) | 27.74 (5.968) | 28.26 (5.672)
Participants with Medical History [Count of Participants; unit: Participants] — Number of participants with at least one clinically relevant medical history/condition (rheumatoid arthritis [RA], ankylosing spondylitis [AS], or psoriatic arthritis [PsA]) were reported.
  Participants | 221 | 107 | 328
Surgery Status [Count of Participants; unit: Participants] — Surgery status was defined as 'yes', if the participant had prior surgical treatment related to the treatment of RA, PsA or AS, and as 'no' if did not have prior surgical treatment.
  Participants
    Yes | 20 | 12 | 32
    No | 201 | 95 | 296

OUTCOME MEASURES:

1. Primary Outcome: Treatment Persistence With CT-P13 in Participants With Rheumatoid Arthritis (RA), Ankylosing Spondylitis (AS) or Psoriatic Arthritis (PsA)
Description: Persistence (in days) was defined as a continuous variable measured in time from index date until date of drug discontinuation. Drug discontinuation was defined as either switching to another non infliximab BDMARD or elapsing of a drug free interval of 16 weeks from CT-P13. For participants undergoing a switch to CT-P13 from Remicade, the index date was considered the date from which Remicade was originally commenced and for participants who initiated treatment with CT-P13 as their first biologic, the index date was considered the date from which CT-P13 was initiated.
Time Frame: During the observation period of 2 years
Population: The safety population was defined as all participants who received at least one dose of CT-P13 during the study observation period.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 221 | 107
days | 404.10 (291.33) | 542.30 (268.55)

2. Primary Outcome: Disease Duration in Participants With Rheumatoid Arthritis (RA), Ankylosing Spondylitis (AS) or Psoriatic Arthritis (PsA), as Recorded on the Day of Inclusion in Study
Description: Disease duration was defined as the number of months from initial diagnosis of rheumatoid disease (RA, AS or PsA) to the date of informed consent, which was recorded at the time of inclusion in the study (Day 1).
Time Frame: At Day 1 of 2 year observation period
Population: The safety population was defined as all participants who received at least one dose of CT-P13 during the study observation period. Here, 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Median (Full Range); unit: months
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 221 | 107
months
  Disease Type: RA: number analyzed (Participants) | 94 | 41
  Disease Type: RA | 52.928 [0.03 to 563.91] | 189.142 [12.65 to 400.20]
  Disease Type: AS: number analyzed (Participants) | 78 | 38
  Disease Type: AS | 35.039 [0.03 to 551.89] | 159.376 [14.65 to 418.33]
  Disease Type: PsA: number analyzed (Participants) | 49 | 28
  Disease Type: PsA | 33.084 [0.03 to 386.50] | 133.979 [18.40 to 464.07]

3. Primary Outcome: Initial Dose of CT-P13 Infusion Administered to Participants
Description: Initial dose of CT-P13 infusion (dose at the time of CT-P13 treatment initiation) was reported in this outcome measure.
Time Frame: At Day 1 of 2 year observation period
Population: The safety population was defined as all participants who received at least one dose of CT-P13 during the study observation period. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: milligram per kilogram
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 207 | 102
milligram per kilogram | 3.00 [2.40 to 6.20] | 4.00 [2.00 to 6.60]

4. Primary Outcome: Number of Participants by Initial Frequency of CT-P13 Infusion Received
Description: Initial frequency of CT-P13 infusion was categorized as: once every 4, 6, 8 weeks and other. 'Other' included all other frequencies other than specified. Number of participants by baseline infusion frequency (in weeks) were reported.
Time Frame: Baseline (Day 1) of 2 year observation period
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 207 | 102
Participants
  Once every 4 weeks | 3 | 1
  Once every 6 weeks | 79 | 42
  Once every 8 weeks | 73 | 44
  Other | 52 | 15

5. Primary Outcome: Total Dose of CT-P13 Infusion Received During Observation Period
Description: Total dose of infusion received by the participants were evaluated.
Time Frame: During the observation period of 2 years
Population: as for outcome 1
Measure: Median (Full Range); unit: milligram per kilogram
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 221 | 107
milligram per kilogram | 35.00 [2.40 to 90.00] | 46.50 [3.00 to 112.20]

6. Primary Outcome: Number of Participants With Change in CT-P13 Infusion Dose
Description: Participants who had change in the dose of infusion (either dose reduction or increase in dose) during the observation period were reported.
Time Frame: During the observation period of 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 221 | 107
Participants | 40 | 8

7. Primary Outcome: Number of Participants Who Had At Least One Concomitant Medication Related to the Treatment of Rheumatoid Arthritis (RA), Ankylosing Spondylitis (AS) or Psoriatic Arthritis (PsA)
Description: Concomitant medications included corticosteroids, non-steroidal anti- inflammatory drugs (NSAID'S) and immunosuppressant. Participants were counted in more than one categories. 'Others' included DMARDS and other medications apart from the categories specified.
Time Frame: During the observation period of 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 221 | 107
Participants
  Corticosteroids | 28 | 2
  NSAID's | 27 | 5
  Immunosuppressants | 48 | 12
  Other | 26 | 2
  Missing | 7 | 5

8. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent were events between first dose of infusion up to 2 years, that were absent before treatment or that worsened relative to pretreatment state. Serious infections including sepsis (excluding opportunistic infections and tuberculosis) were the pre-defined TEAE of special Interest for this study. AEs included both serious and non-serious adverse events.
Time Frame: During the observation period of 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 221 | 107
Participants
  TEAEs | 97 | 29
  SAEs | 19 | 10
  TEAEs of Special Interest | 24 | 8

9. Secondary Outcome: Change From Baseline in Disease Activity Score-28 (DAS28) in Participants With Rheumatoid Arthritis (RA) at Months 6, 12, 18 and 24
Description: DAS28 calculated from the number of tender joint count (TJC) and swollen joint count (SJC) using 28 joints count, erythrocyte sedimentation rate (ESR) (millimeters per hour; ranged from 0 to 150), and a participant's general health assessment (GH) on a 100 millimeter (mm) visual analog scale (VAS) (ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicated worsening of health condition). Total DAS28 score ranged from 0 (none) to 9.4 (extreme disease activity), higher scores indicated more disease activity. DAS28 less than or equal to (<=) 3.2 implied low, greater than (>) 3.2 to <=5.1 implied moderate, and >5.1 implied high disease activity. DAS28=0.56*sqrt(28TJC)+0.28*sqrt(28SJC)+0.70*ln(ESR)+0.014*GH; where ln = natural logarithm and sqrt = square root of.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: Analysis performed on participants who had received at least one dose of CT-P13 and had at least one post-dose assessment for DAS28. 'Overall number of participants analyzed': participants who were evaluable for this outcome measure. 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 92 | 41
units on a scale
  Baseline: number analyzed (Participants) | 43 | 31
  Baseline | 4.033 (1.5186) | 2.641 (1.1401)
  Change at Month 6: number analyzed (Participants) | 22 | 23
  Change at Month 6 | -1.269 (1.5981) | 0.210 (1.1452)
  Change at Month 12: number analyzed (Participants) | 14 | 14
  Change at Month 12 | -0.642 (1.1220) | -0.432 (1.6097)
  Change at Month 18: number analyzed (Participants) | 1 | 5
  Change at Month 18 | -0.795 | 0.534 (0.9656)
  Change at Month 24: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change From Baseline in Disease Activity Score-28 (DAS28) in Participants With Psoriatic Arthritis (PsA) at Months 6, 12, 18 and 24
Description: DAS28 calculated from the number of TJC and SJC using 28 joints count, ESR (millimeters per hour; ranged from 0 to 150), and participant's GH on a 100 mm VAS (ranging from 0 mm [very well] to 100 mm [extremely bad], higher scores indicated worsening of health condition). Total DAS28 score ranged from 0 (none) to 9.4 (extreme disease activity), higher scores indicated more disease activity. DAS28 <= 3.2 implied low, > 3.2 to <=5.1 implied moderate, and >5.1 implied high disease activity. DAS28=0.56*sqrt(28TJC)+0.28*sqrt(28SJC)+0.70*ln(ESR)+0.014*GH; where ln = natural logarithm and sqrt = square root of.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 46 | 28
units on a scale
  Baseline: number analyzed (Participants) | 22 | 14
  Baseline | 3.755 (1.7767) | 2.351 (1.0677)
  Change at Month 6: number analyzed (Participants) | 13 | 10
  Change at Month 6 | -0.913 (1.8785) | 0.152 (0.2737)
  Change at Month 12: number analyzed (Participants) | 4 | 8
  Change at Month 12 | -0.006 (1.7984) | 0.259 (0.3916)
  Change at Month 18: number analyzed (Participants) | 4 | 4
  Change at Month 18 | -0.747 (1.2115) | 0.840 (0.9880)
  Change at Month 24: number analyzed (Participants) | 1 | 3
  Change at Month 24 | -0.543 | 0.313 (0.2436)

11. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in Participants With Ankylosing Spondylitis (AS) at Months 6, 12, 18 and 24
Description: BASDAI is a self-reported measure of disease activity in participants with AS. Participants answered 6 questions measuring symptoms of AS (fatigue, spinal pain, joint pain or swelling, areas of localized tenderness, morning stiffness duration and severity). The BASDAI total score was calculated by computing the mean of questions 5 and 6 and adding it to the sum of questions (Q) 1-4. This score was then divided by 5. BASDAI=Q1+Q2+Q3+Q4+[Q5+Q6/2]/5. The total BASDAI score ranges from 1=none to 10=severe, where lower score indicated less disease activity. The level of AS disease activity was interpreted as low (BASDAI < 4) or high (BASDAI > 4).
Time Frame: Baseline, Weeks 6, 12, 18 and 24
Population: Analysis performed on participants who had received at least one dose of CT-P13 and had at least one post-dose assessment for BASDAI. 'Overall number of participants analyzed': participants who were evaluable for this outcome measure. 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 77 | 38
units on a scale
  Baseline: number analyzed (Participants) | 65 | 29
  Baseline | 4.63 (2.263) | 3.06 (2.313)
  Change at Month 6: number analyzed (Participants) | 58 | 27
  Change at Month 6 | -1.00 (1.911) | 0.01 (1.470)
  Change at Month 12: number analyzed (Participants) | 36 | 17
  Change at Month 12 | -0.87 (1.816) | 0.06 (2.304)
  Change at Month 18: number analyzed (Participants) | 30 | 11
  Change at Month 18 | -0.55 (2.153) | -0.24 (2.015)
  Change at Month 24: number analyzed (Participants) | 11 | 6
  Change at Month 24 | -1.14 (2.167) | -1.32 (2.875)

12. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) in Participants With Ankylosing Spondylitis (AS) at Months 6,12,18 and 24
Description: ASDAS is used to assess disease activity in participants with AS. It is a score combining the assessment of overall pain (Q1), duration of morning stiffness (Q2), peripheral pain/swelling (Q3), PtGA (assessed on a sale of 0 to 10, where 0 = not active and 10=very active), and C-reactive protein (CRP) in milligrams per liter (mg/L). ASDAS total score was derived using the following formula: ASDAS=0.12*Q1+0.06*Q2+0.11*GH+0.07*Q3+0.58*ln (CRP+1). The level of AS disease activity was interpreted as inactive disease (ASDAS< 1.3), moderate disease activity (1.3 <= ASDAS < 2.1), high disease activity (2.1<= ASDAS <=3.5) and very high disease activity (ASDAS > 3.5).
Time Frame: Baseline, Weeks 6, 12, 18 and 24
Population: Analysis performed on participants who had received at least one dose of CT-P13 and had at least one post-dose assessment for ASDAS. 'Overall number of participants analyzed': participants who were evaluable for this outcome measure. 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 77 | 38
units on a scale
  Baseline: number analyzed (Participants) | 32 | 16
  Baseline | 3.153 (1.1082) | 2.151 (1.0456)
  Change at Month 6: number analyzed (Participants) | 18 | 13
  Change at Month 6 | -0.875 (1.3108) | -0.023 (1.1017)
  Change at Month 12: number analyzed (Participants) | 16 | 9
  Change at Month 12 | -0.379 (0.9905) | -0.452 (0.8156)
  Change at Month 18: number analyzed (Participants) | 6 | 3
  Change at Month 18 | -0.603 (2.7745) | -0.002 (0.3630)
  Change at Month 24: number analyzed (Participants) | 6 | 4
  Change at Month 24 | -1.154 (1.2293) | -0.356 (1.7080)

13. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) in Participants With Ankylosing Spondylitis (AS) at Months 6, 12, 18 and 24
Description: BASFI is a validated self assessment tool to determine the degree of functional limitation in participants with AS. It is comprised of 10 questions which were answered by participants using a VAS ranging from 0 (being easy) to 10 (impossible). BASFI total score was calculated as the average score of the 10 questions, and ranges from 0 (no functional impairment) to 10 (maximal impairment), higher scores indicated more impairment.
Time Frame: Baseline, Weeks 6, 12, 18 and 24
Population: Analysis performed on participants who had received at least one dose of CT-P13 and had at least one post-dose assessment for BASFI. 'Overall number of participants analyzed': participants who were evaluable for this outcome measure. 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 77 | 38
units on a scale
  Baseline: number analyzed (Participants) | 63 | 29
  Baseline | 4.17 (2.804) | 2.89 (2.492)
  Change at Month 6: number analyzed (Participants) | 57 | 27
  Change at Month 6 | -0.72 (2.107) | 0.20 (1.146)
  Change at Month 12: number analyzed (Participants) | 35 | 17
  Change at Month 12 | -1.01 (2.085) | 0.18 (2.228)
  Change at Month 18: number analyzed (Participants) | 29 | 11
  Change at Month 18 | -0.43 (2.194) | 0.23 (2.257)
  Change at Month 24: number analyzed (Participants) | 11 | 6
  Change at Month 24 | -1.18 (2.379) | -0.42 (3.012)

14. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score at Months 6, 12, 18 and 24
Description: HAQ-DI assesses the degree of difficulty a participant had experienced in 8 domains of daily activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip and other activities. Each item scored on a 4-point scale from 0 to 3 with 0 ="no difficulty", 1 ="some difficulty", 2 = "much difficulty", and 3 ="unable to do". Overall score was computed as the sum of scores divided by the number of domains answered. Total possible score range was 0-3 with 0 = "no difficulty to 3 ="unable to do". Higher score indicate more difficulty in performing daily living activities.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: Analysis performed on participants who had received at least one dose of CT-P13 during the study observation period and had at least one post-dose assessment of HAQ-DI. Here 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 215 | 107
units on a scale
  Baseline: number analyzed (Participants) | 181 | 85
  Baseline | 0.956 (0.7493) | 0.646 (0.6684)
  Change at Month 6: number analyzed (Participants) | 162 | 76
  Change at Month 6 | -0.216 (0.5906) | 0.026 (0.3648)
  Change at Month 12: number analyzed (Participants) | 90 | 52
  Change at Month 12 | -0.207 (0.5739) | -0.043 (0.5144)
  Change at Month 18: number analyzed (Participants) | 75 | 24
  Change at Month 18 | -0.150 (0.4650) | -0.021 (0.3878)
  Change at Month 24: number analyzed (Participants) | 22 | 9
  Change at Month 24 | -0.398 (0.6918) | -0.153 (0.7336)

15. Secondary Outcome: Change From Baseline in European Quality of Life- 5 Dimensions 3 Level Version (EQ-5D-3L) Visual Analog Scale (VAS) Score at Months 6, 12, 18 and 24
Description: EQ-5D-3L is a standardized, participant-administered measure of health outcomes. It consists of two parts: EQ-5D descriptive system (Part I) and the EQ-VAS (Part II). EQ-5D-3L Part II uses a vertical graduated VAS to measure health status on a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicating a better health state.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: Analysis was performed on participants who had received at least one dose of CT-P13 during the study observation period and had at least one post-dose assessment of EQ-5D-3L. Here 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 215 | 107
units on a scale
  Baseline: number analyzed (Participants) | 183 | 85
  Baseline | 62.7 (23.55) | 70.0 (22.71)
  Change at Month 6: number analyzed (Participants) | 163 | 76
  Change at Month 6 | 6.0 (25.55) | 0.2 (20.66)
  Change at Month 12: number analyzed (Participants) | 87 | 52
  Change at Month 12 | 4.2 (21.93) | 1.0 (26.06)
  Change at Month 18: number analyzed (Participants) | 75 | 24
  Change at Month 18 | -0.8 (28.71) | -0.0 (25.98)
  Change at Month 24: number analyzed (Participants) | 21 | 9
  Change at Month 24 | 4.3 (16.28) | 12.4 (30.99)

16. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-3 Levels (EQ-5D-3L) Index Score at Months 6, 12, 18 and 24
Description: EQ-5D-3L is a standardized, participant-administered measure of self-reported health outcomes. It consists of two parts: EQ-5D descriptive system (Part I) and the EQ-VAS (Part II). For Part I, i.e. EQ-5D-3L index score, participants rated their current health state on 5 single-item dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with each dimension having three levels of function:. 1=no problems, 2=some problems and 3=extreme problems. Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score was transformed and results in a total score range of -0.074 to 1.00; higher scores indicating a better health state.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 215 | 107
units on a scale
  Baseline: number analyzed (Participants) | 183 | 85
  Baseline | 0.627 (0.2260) | 0.757 (0.1906)
  Change at Month 6: number analyzed (Participants) | 163 | 76
  Change at Month 6 | 0.097 (0.2309) | 0.004 (0.1859)
  Change at Month 12: number analyzed (Participants) | 87 | 52
  Change at Month 12 | 0.106 (0.2093) | -0.002 (0.1900)
  Change at Month 18: number analyzed (Participants) | 75 | 24
  Change at Month 18 | 0.102 (0.1522) | -0.041 (0.1416)
  Change at Month 24: number analyzed (Participants) | 21 | 9
  Change at Month 24 | 0.090 (0.1479) | -0.004 (0.1735)

17. Secondary Outcome: Change From Baseline in Physical Component Summary (PCS) Score of Short Form 12 Version 2 (SF-12v2) Health Survey at Months 6, 12, 18 and 24
Description: The SF-12v2 is a self-administered, validated, multipurpose SF questionnaire to measure generic health status. It consists of 12 items, which are categorized into eight domains (subscales) of functioning and well-being: physical function, role limitations due to physical problems, bodily pain, general health perceptions, energy and vitality, social functioning, role limitations due to emotional problems, and mental health. The score range for each of the 8 health aspects was from 0 (poor health) to 100 (better health), higher scores indicating good health condition. These eight domains are further summarized into PCS and mental component summary (MCS). The score range for each of these 2 summary scores was from 0 (poor health) to 100 (better health). Higher scores indicated a better health-related quality of life.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: Analysis was performed on participants who had received at least one dose of CT-P13 during the study observation period and had at least one post-dose assessment of SF-12v2. Here 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 215 | 107
units on a scale
  Baseline: number analyzed (Participants) | 181 | 85
  Baseline | 37.018 (10.1214) | 41.865 (10.2835)
  Change at Month 6: number analyzed (Participants) | 162 | 76
  Change at Month 6 | 2.679 (9.5359) | 0.638 (7.5793)
  Change at Month 12: number analyzed (Participants) | 90 | 52
  Change at Month 12 | 3.988 (8.6626) | 0.683 (8.8907)
  Change at Month 18: number analyzed (Participants) | 75 | 24
  Change at Month 18 | 2.325 (8.1633) | 0.295 (11.0411)
  Change at Month 24: number analyzed (Participants) | 22 | 9
  Change at Month 24 | 4.238 (9.2347) | 1.712 (7.9035)

18. Secondary Outcome: Change From Baseline in Mental Component Summary (MCS) Score of Short Form 12 Version 2 (SF-12v2) Health Survey at Months 6, 12, 18 and 24
Description: as for outcome 17
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 215 | 107
units on a scale
  Baseline: number analyzed (Participants) | 181 | 85
  Baseline | 47.154 (10.9659) | 52.152 (9.8788)
  Change at Month 6: number analyzed (Participants) | 162 | 76
  Change at Month 6 | 2.603 (8.9694) | -0.412 (8.7364)
  Change at Month 12: number analyzed (Participants) | 90 | 52
  Change at Month 12 | 1.435 (8.1599) | 0.119 (8.3434)
  Change at Month 18: number analyzed (Participants) | 75 | 24
  Change at Month 18 | 1.457 (8.0383) | -1.145 (9.9283)
  Change at Month 24: number analyzed (Participants) | 22 | 9
  Change at Month 24 | -0.593 (9.7558) | 5.111 (5.0804)

19. Secondary Outcome: Change From Baseline in Physician Global Assessment (PGA) of Rheumatoid Diseases Activity at Months 6, 12, 18 and 24
Description: PGA of disease activity was measured on a 0 to 100 mm VAS, where 0 mm = no disease activity and 100 mm = extremely active. Higher scores indicated worsening of condition.
Time Frame: Baseline, Months 6, 12, 18 and 24
Population: Analysis was performed on participants who had received at least one dose of CT-P13 during the study observation period and had at least one post-dose assessment of PGA. Here 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
Number analyzed (Participants) | 215 | 107
millimeters
  Baseline: number analyzed (Participants) | 176 | 88
  Baseline | 34.9 (27.80) | 18.4 (17.27)
  Change at Month 6: number analyzed (Participants) | 159 | 74
  Change at Month 6 | -13.4 (26.94) | 0.6 (18.07)
  Change at Month 12: number analyzed (Participants) | 91 | 50
  Change at Month 12 | -19.2 (23.17) | -1.5 (19.02)
  Change at Month 18: number analyzed (Participants) | 66 | 26
  Change at Month 18 | -12.5 (20.58) | 2.1 (11.75)
  Change at Month 24: number analyzed (Participants) | 18 | 11
  Change at Month 24 | -25.6 (23.49) | -3.4 (12.27)

ADVERSE EVENTS:
Time Frame: During the observation period of 2 years
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population was evaluated.
Arm/Group | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive | Participants Who Switched From Remicade to CT-P13
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/107
Serious Adverse Events (participants affected / at risk) | 19/221 | 10/107
Other Adverse Events (participants affected / at risk) | 88/221 | 24/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive (N=221) | Participants Who Switched From Remicade to CT-P13 (N=107)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Necrotising herpetic retinopathy (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Device loosening (Product Issues) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Biologic Disease Modifying Anti-Rheumatic Drugs (BDMARD) Naive (N=221) | Participants Who Switched From Remicade to CT-P13 (N=107)
Cardiomyopathy (Cardiac disorders) | 1 | 0
Uveitis (Eye disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Cyst (General disorders) | 0 | 1
Drug ineffective (General disorders) | 25 | 6
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Nodule (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 0
Cystitis (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Nasal herpes (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 6 | 1
Oral herpes (Infections and infestations) | 0 | 2
Periodontitis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 4
Urinary tract infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0
Exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 14 | 2
Blood pressure increased (Investigations) | 1 | 0
Drug specific antibody (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Mycobacterium tuberculosis complex test positive (Investigations) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 6 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Palmoplantar pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
Carpal tunnel decompression (Surgical and medical procedures) | 1 | 0
Varicose vein operation (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Due to erroneous data transmission/ data discrepancies which occurred with use of the electronic data capture tool, data summaries only for a portion of the data for OM 9 to 19, which corresponded to visit dates in clinical database were provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-05-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT02605642/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT02605642/SAP_001.pdf